CLINICAL TRIAL: NCT07372690
Title: Using Goal Attainment Scale (GAS) to Increase Active Involvement of Patients and Their Family in the Identification of Functional Objectives During Hospitalization for Hematopoietic Stem Cell Transplantation (HSCT): a Randomized Controlled Trial.
Brief Title: Goal Attainment Scale in Transplantation
Acronym: GAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Full Professor, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GAST; 137/2022 (Other: Comitato Etico Interaziendale AOU Città della Salute e della Scienza di Torino, AO Mauriziano e ASL Città di Torino)
Record Dates: First submitted 2025-12-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Oncology; Hematology
Keywords: adolescents; children; hematopoietic stem cell transplantation; physical therapy; motor performance; fatigue; family centered care
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise programme (EP) and rehabilitation counselling indication (RCI) (Other): Exercise Program EP is carried out five days a week (two days independently with parental support and three days under supervision). Each 30-minute session is supervised by one therapist for all patients. The EP programme includes three types of exercise: muscle-strengthening exercises for the upper and lower extremities, preceded by a 10-minute warm-up; 15 minutes of aerobic exercise; and 5 minutes of stretching.
  Rehabilitation counselling indications RCI have to be followed daily. RCI consist of some practical advice on how to adopt an active lifestyle during recovery. Some examples are getting up to go to the bathroom or the window to talk to visitors, sitting on a chair for school lessons.
  Interventions: Other: control group
- Exercise programme (EP), rehabilitation counselling indication (RCI) and Goal Attaiment Scale (GAS) (Experimental): Exercise Program EP is carried out five days a week (two days independently with parental support and three days under supervision). Each 30-minute session is supervised by one therapist for all patients. The EP programme includes three types of exercise: muscle-strengthening exercises for the upper and lower extremities, preceded by a 10-minute warm-up; 15 minutes of aerobic exercise; and 5 minutes of stretching.
  Rehabilitation counselling indications RCI have to be followed daily. RCI consist of some practical advice on how to adopt an active lifestyle during recovery. Some examples are getting up to go to the bathroom or the window to talk to visitors, sitting on a chair for school lessons.
  GAS During their hospitalisation, children and caregivers in the experimental group define a functional goal together each week with the help of the therapist. This is verified using Goal Attainment Scaling, which identifies specific and significant objectives for the patient and their family.
  Interventions: Other: GAS group

INTERVENTIONS:
Other: GAS group — This intervention includes an exercise programme (EP) and rehabilitation counselling indication (RCI) during hospitalisation for HSCT. Participants in the experimental group also set their own functional goals using GAS (Goal Attainment Scaling) with the help of the therapist during hospitalization.
  EP is carried out five days/week (30-minute per session) and it consists in muscle-strengthening, aerobic and stretching exercises.
  RCI have to be followed daily and they are some practical advice on how to adopt an active lifestyle during recovery.
  GAS is structured around the definition of a starting level (-1) and the goal to be achieved (level 0). Two higher levels (+1 and +2) are used to indicate better performance than expected, and level -2 is used to indicate regression in the initial functional objective. The "Goaled" app, which is available for free on smartphones and tablets, is used to define and verify the objectives. This should increase patient's motivation.
  Arms: Exercise programme (EP), rehabilitation counselling indication (RCI) and Goal Attaiment Scale (GAS)
Other: control group — Participants assigned in this group follow an Exercise Program and Rehabilitation counselling indications.
  Exercise Program EP is carried out five days a week (two days independently with parental support and three days under supervision). Each 30-minute session is supervised by one therapist for all patients. The EP programme includes three types of exercise: muscle-strengthening exercises for the upper and lower extremities, preceded by a 10-minute warm-up; 15 minutes of aerobic exercise; and 5 minutes of stretching.
  Rehabilitation counselling indications RCI have to be followed daily. RCI consist of some practical advice on how to adopt an active lifestyle during recovery. Some examples are getting up to go to the bathroom or the window to talk to visitors, sitting on a chair for school lessons.
  Arms: Exercise programme (EP) and rehabilitation counselling indication (RCI)

SUMMARY:
The primary aim of this monocentric randomised controlled study is to evaluate the impact of using GAS to maintain the functional abilities of children and adolescents undergoing TCSE. The secondary aims include evaluating parents' and adolescents' perceived changes in the subject's functional abilities from the moment of stem cell transplantation unit (SCTU) admission to subsequent follow-ups. Another secondary aim is to evaluate the achievement of functional goals as defined by GAS in the experimental group (EG). Other aims include investigating the feasibility of the exercise program and the rehabilitation counselling indications in both groups, as well as the effectiveness of the two interventions and GAS use in the EG.

DETAILED DESCRIPTION:
HSCT is a potentially curative option for many diseases, including haematological malignancies and refractory solid tumours in children and adolescents. Its use in this age group has increased over the last three decades, as have survival rates decades. However, HSCT can cause a significant number of clinical complications and side effects in both the short and long term. Short-term effects include mucositis, fever, nausea and vomiting, while long-term effects include organ toxicity and fatigue. Allogeneic HSCT recipients can indeed develop graft-versus-host disease, which can lead to extensive multiorgan failure, systemic toxicity and mortality. Previous treatments, the severity of the conditioning regimen, the length of isolation and hospitalisation can all severely impair physical, cognitive and psychosocial functions, resulting in a reduction in quality of life (QoL). Recent studies have shown that exercise and rehabilitation are promising tools for decreasing the side effects of HSCT and improving QoL in the paediatric population undergoing HSCT). A systematic meta-analysis review reported that physical exercise is safe, feasible, and effective in preventing the decline in quality of life and physical performance in paediatric patients undergoing HSCT.

It is widely recognized that rehabilitation treatment in developmental age should consider the multiplicity of altered motor, perceptive, cognitive, affective, communicative and relational functions, their mutual interactions, as well as variables such as age and the role of the family, while respecting the individuality of each child. Health care professionals should treat patients with dignity, sensitivity, kindness, and respect for their individual needs and preferences for medical, clinical and rehabilitative care. These principles characterize the Family Centered Care (FCC), an approach based on the active involvement of the patients and their families in the care process. Other studies showed that uptake of an FCC approach in paediatric settings can positively impact children's HRQL. The FCC approach has been recognized as a model of best practice in pediatric rehabilitation, where it can be integrated in the rehabilitation programme by identifying clinically relevant and functional goals for the patients and their caregivers. Moreover, the approach can increase patient's compliance. Goal Attainment Scaling (GAS) has revealed itself as being a powerful tool to establish personalized goals and to objectively quantify the benefits of rehabilitation treatment. The GAS value lies in the possibility of identifying specific concrete objectives for each patient. The tool, which is used in different fields, is widely applied in pediatric rehabilitation. To date, the effects of active involvement of children, adolescents and their families in the definition of functional goals during hospitalization for HSCT have not yet been studied. The use of GAS to identify and achieve personalized, concrete and functional short-term goals during hospitalization could help patients to maintain a more active lifestyle. Consequently, it will reduce sedentary behaviors which are very frequent in this population. The increase in activity levels could significantly contribute to the maintenance of functional abilities that are often reduced during the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 months - 17 years and 11 months
* diagnosis of oncological or hematological disease undergoing HSCT
* No specific rehabilitation treatment ongoing at the moment of recruitment
* Written informed consent from patient or parents/legal representative, and age-appropriate assent.

Exclusion Criteria:

* Patients that are not able and willing to comply with study visits and procedures.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-12-23 (Estimated)

PRIMARY OUTCOMES:
Functional Abilities Assessment in Paediatric Oncology (FAAPO) Scale | - At the admission to the ward - At hospital discharge - At 60 days after HSCT
  This tool is a short version of the Gross Motor Function Measure and has been validated for use with Italian paediatric oncology patients aged 6 months to 18 years. It comprises 36 items, each of which can be scored as 0, 1, 2, 3 or 'not tested'. The scoring key is as follows: 0 - does not initiate; 1 - initiates; 2 - partially completes; and 3 - completes. The final FAAP-O score provides a percentage of functional abilities.

SECONDARY OUTCOMES:
Global Rating of Change (GCR) | - At hospital discharge - At 60 days after HSCT
  Change in functional abilities perceived by parents and adolescents between T0 and T1, and between T1 and T2, is tested using Global Rating of Change (GCR).
Achievement of the functional objectives established with GAS (Goal Attainment Scaling) | Each 7 days from the baseline to the discharge from the ward.
  Achievement of the functional objectives established with GAS in the experimental group, using GAS.
Percentage of adherence to the exercise programme and rehabilitation counselling indications. | Each 7 days from the baseline to the discharge from the ward.
  Percentage of adherence to the exercise programme and rehabilitation counselling indications.
Percentage of GAS application in the experimental group. | Each 7 days from the baseline to the discharge from the ward.
  Percentage of GAS application in the experimental group.
Sit and Reach Test | - At the admission to the ward - At hospital discharge - At 60 days after HSCT
  Muscle extensibility of the posterior kinetic chain is measured with Sit and Reach Test. It is performed by sitting with legs extended against a box, then reaching forward as far as possible over the measuring line, holding for 2 seconds. It's scored by measuring the distance fingertips reach past (positive) or short of (negative) the toes.
Hand grip test | - At the admission to the ward - At hospital discharge - At 60 days after HSCT
  The Hand Grip Test measures maximum isometric hand and forearm strength using a dynamometer, assessing overall physical capacity and potential indicators of health, functional status, and malnutrition. The procedure consists in squeezing the device for a few seconds, recording the force (in lbs), and often repeating trials to find the best score.
Time Up and Go Test | - At the admission to the ward - At hospital discharge - At 60 days after HSCT
  The Timed Up and Go (TUG) test is a functional mobility assessment test. It requires a chair, stopwatch, and tape to mark 3 meters. A person stands from the chair, walks to the line at a normal pace, turns, walks back, and sits down, with the time recorded from "go" until seated.
2-Minutes Walking Test | - At the admission to the ward - At hospital discharge - At 60 days after HSCT
  The 2-Minute Walk Test (2MWT) assesses a person's walking endurance and aerobic capacity. It is measured with the maximum distance they can cover in two minutes, walking back and forth along a clear, standardized path (30 metres), at their fastest safe pace.
Pediatric Quality of Life Multidimensional Fatigue Scale | - At the admission to the ward - At 60 days after HSCT
  The Pediatric Quality of Life Multidimensional Fatigue Scale (PedsQL - MFS) is an 18-item questionnaire from the Pediatric Quality of Life Inventory (PedsQL) used to measure fatigue in children and adolescents (ages 2-18), assessing three specific dimensions: General Fatigue, Sleep/Rest Fatigue, and Cognitive Fatigue, with higher scores indicating better quality of life and less fatigue, using a Likert-type scale from "never" to "almost always". e;
Pediatric Quality of Life Cancer Module | - At the admission to the ward - At 60 days after HSCT
  The Pediatric Quality of Life Cancer Module (PedsQL Cancer Module) is a widely used, cancer-specific questionnaire measuring health-related quality of life (HRQoL) in children and adolescents with cancer, using both child self-report and parent proxy-report, assessing dimensions like pain, fatigue, treatment anxiety, and appearance.
Changes in immunological variables | - At 60 days after HSCT - At 90 days after HSCT
  Immune recovery will be evaluated through the counting of the different populations of white blood cells (leukocytes, monocytes and lymphocytes), of the lymphocyte subpopulations (total T lymphocytes (CD45+ CD3+ CD56-), B lymphocytes (CD19+ CD20+), NK lymphocytes (CD45+ CD3- CD56+), CD4+ T lymphocytes (CD3+ CD4+ CD8-) and CD8+ T lymphocytes (CD3+ CD4- CD8 +).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Saglio, PhD Medical Doctor, Principal Investigator — A.O.U. Città della Salute e della Scienza - OIRM
Locations (1):
- A.O.U. Città della Salute e della Scienza - OIRM, Torino, TO, Italy